CLINICAL TRIAL: NCT01647958
Title: Transoral Incisionless Fundoplication (TIF) Versus Medical Proton Pump Inhibitor (PPI) Management of Refractory Gastroesophageal Reflux Disease (GERD) Symptoms
Brief Title: The EndoGastric Solutions TEMPO Trial
Acronym: TEMPO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: EndoGastric Solutions (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: D01292
Record Dates: First submitted 2012-06-22; First posted 2012-07-24 (Estimated); Results first posted 2020-11-02 (Actual); Last update posted 2020-11-23 (Actual); Status verified 2020-11

CONDITIONS: Gastroesophageal Reflux Disease (GERD)
Keywords: TEMPO; TIF; Transoral Incisionless Fundoplication; EsophyX System; refractory symptoms; proton pump inhibitors; EndoGastric Solutions; EGS; Acid Reflux; Heartburn; Regurgitation
MeSH Terms: conditions — Gastroesophageal Reflux; Heartburn

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment Arm (Experimental): Transoral incisionless esophago-gastric fundoplication using the EsophyX system with SerosaFuse fasteners (EndoGastric Solutions, Inc., Redmond, WA, USA) and following TIF2.0 protocol.
  Interventions: Device: EsophyX System with SerosaFuse fasteners
- Control (Active Comparator): Patients who are dependent upon daily PPIs will continue on single dose twice daily or increase to single dose twice daily for the first six months of the clinical trial. Patients will be offered TIF crossover procedure upon completion of month-6 follow-up visit.
  Interventions: Drug: PPI

INTERVENTIONS:
Device: EsophyX System with SerosaFuse fasteners — Transoral Incisionless Fundoplication (TIF)/Transoral incisionless esophago-gastric fundoplication using the EsophyX System with SerosaFuse fasteners
  Arms: Treatment Arm
Drug: PPI — Control Arm participants will take maximum standard dose of PPI during Initial Study period
  Other Names: same brand of PPI used by all Control Arm participants
  Arms: Control

SUMMARY:
The purpose of this study is to assess the efficacy and safety of Transoral Incisionless Fundoplication (TIF) performed with EsophyX as compared to proton pump inhibitor (PPI) therapy for the treatment of chronic Gastroesophageal Reflux Disease (GERD) patients with refractory symptoms on Proton Pump Inhibitors (PPIs).

DETAILED DESCRIPTION:
The objective of this study is to assess the efficacy and safety of TIF performed with EsophyX as compared to proton pump inhibitor (PPI) therapy for the treatment of chronic GERD patients with medically refractory GERD symptoms other than heartburn.

Primary hypothesis: TIF will be superior to PPIs in eliminating or significantly improving daily bothersome GERD symptoms and/or troublesome regurgitation, if present, at 6-month follow-up. Secondary hypotheses: TIF will be superior to PPIs in eliminating or significantly improving daily bothersome GERD symptoms and/or troublesome regurgitation, if present, at 12-, 24-, 36-, 48- and 60-month follow-up. The majority of surgical patients will have normalized or 50% improved esophageal acid exposure compared to baseline at 6-month follow-up. The majority of surgical patients will be completely off PPIs at 6-, 12-, 24-, 36-, 48- and 60-month follow-up compared to baseline. The majority of crossover patients will be completely off PPIs at 6-, 18-, 30-, 42- and 54-month follow-up compared to baseline. A statistically greater proportion of crossover patients treated with TIF will be free of daily bothersome symptom(s) or will experience clinically significant improvement at 6-, 18-, 30-, 42- and 54-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-80 years;
2. GERD for > 1 year;
3. History of daily PPIs for > 6 months;
4. At least daily bothersome medically refractory GERD symptom(s) other than heartburn on PPIs;
5. Hill grade I and II at gastroesophageal junction;
6. Proven gastroesophageal reflux by either endoscopy, ambulatory pH or barium swallow testing;
7. Willingness to undergo pH testing;
8. Willingness to cooperate with the postoperative diet;
9. Availability for follow-up visits at 6, 12, 24, and 36 months;
10. Willingly and cognitively signed inform consent

Exclusion Criteria:

1. BMI > 35 Hiatal hernia > 2c m in axial height and > 2 cm in greatest transverse dimension;
2. Esophagitis grade C and D;
3. Barrett's esophagus > 2 cm;
4. Esophageal ulcer;
5. Fixed esophageal stricture or narrowing;
6. Portal hypertension and/or varices;
7. Active gastro-duodenal ulcer disease; Gastric outlet obstruction or stenosis;
8. Gastroparesis;
9. Coagulation disorders;
10. History of any of the following: resective gastric or esophageal surgery, antireflux surgery with anatomy unsuitable for TIF procedure per physician judgment, cervical spine fusion, Zenker's diverticulum, esophageal epiphrenic diverticulum, achalasia, scleroderma or dermatomyositis, eosinophilic esophagitis, or cirrhosis;
11. Pregnancy or plans of pregnancy in the next 12 months;
12. Enrollment in another device or drug study that may confound the results

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2012-06-01 (Actual); Primary Completion 2015-10-01 (Actual); Study Completion 2017-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karim Trad, MD, FACS, Principal Investigator — Reston Surgical Associates
Locations (1):
- EndoGastric Solutions, Redmond, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Trad KS, Simoni G, Barnes WE, Shughoury AB, Raza M, Heise JA, Turgeon DG, Fox MA, Mavrelis PG. Efficacy of transoral fundoplication for treatment of chronic gastroesophageal reflux disease incompletely controlled with high-dose proton-pump inhibitors therapy: a randomized, multicenter, open label, crossover study. BMC Gastroenterol. 2014 Oct 6;14:174. doi: 10.1186/1471-230X-14-174. PMID 25284142
- See also: EndoGastric Solutions Company Page — http://www.endogastricsolutions.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from seven U.S. hospitals.
Pre-assignment Details: 65 patients randomized: 41 treatment, 24 control. 39 and 21 respectively, were completed. Control-arm patients offered Crossover to TIF following 6 mo. follow-up visit. 21 control-arm patients crossed over to TIF procedure after 6-month follow-up. Note: 6 mo. difference between Crossover and Treatment patient post-hoc results. Extended Results Phase (3 and 5yr follow-up) participants are placed in a single cohort of Treatment + Control arm patients.
Groups:
- Treatment Arm: Transoral incisionless esophago-gastric fundoplication using the EsophyX system with SerosaFuse fasteners (EndoGastric Solutions, Inc., Redmond, WA, USA) and following TIF2.0 protocol.
  EsophyX System with SerosaFuse fasteners: Transoral Incisionless Fundoplication (TIF)/Transoral Incisionless Esophago-Gastric Fundoplication
- Control: Patients who are dependent upon daily PPIs will continue on single dose twice daily or increase to single dose twice daily for the first six months of the clinical trial.
Period: Initial Study
Arm/Group | Treatment Arm | Control
Started | 41 | 24
Completed | 39 | 21
Not Completed | 2 | 3
Not completed — Lost to Follow-up | 2 | 3
Period: Continuation Phase
Arm/Group | Treatment Arm | Control
Started | 39 | 21
Completed | 0 (Treatment-arm patients received TIF procedure during Initial Study phase) | 21 (21 Control patients received TIF crossover procedure following 6-month follow-up visit.)
Not Completed | 39 | 0
Not completed — treatment received during Overall Study | 39 | 0
Period: Extended Follow-up Phase
Arm/Group | Treatment Arm | Control
Started | 60 (Treatment and Control/Crossover patients were combined into 1 cohort for this follow up. 39+21=60) | 0 (Treatment and Control/Crossover patients combined into 1 cohort for this period=60, 0 under Control)
Completed | 52 (The 8 lost to follow up patients are of the combined Treatment and Control cohort of 52 patients) | 0
Not Completed | 8 | 0
Not completed — Lost to Follow-up | 8 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Arm | Control | Total
Number analyzed (Participants) | 39 | 21 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 34 | 21 | 55
  >=65 years | 5 | 0 | 5
Age, Continuous [Median (Full Range); unit: years] | 54.8 [35.7 to 73.3] | 50.1 [32.5 to 63.3] | 53.16 [32.5 to 73.3]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 13 | 33
  Male | 19 | 8 | 27
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 39 | 21 | 60

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting GERD (Gastroesophageal Reflux Disease) Symptom Elimination or Clinically Significant Improvement Evaluated by RSI (Reflux Symptom Index) and RDQ (Reflux Disease Questionnaire).
Description: Elimination or clinically significant improvement in GERD symptoms, other than heartburn, refractory to PPI, evaluated by Reflux Symptom Index (RSI):9-item questionnaire measures atypical symptoms: hoarseness, throat clearing, excess throat mucus, dysphagia, cough. Scale for each item ranges from 0 (no problem) to 5 (severe), with max total score of 45, normality threshold of ≤13. Reflux Disease Questionnaire (RDQ):12-item questionnaire to assess frequency and severity of heartburn (4 items measure frequency/severity of pain and burning behind breastbone), regurgitation (4 items measure frequency/severity of acid taste in mouth and movement of material upward from stomach), and dyspeptic complaints (4 items measure frequency and severity of pain or burning in upper stomach). Responses from 0 (not present) to 5 (daily) for frequency and 0 (not present) to 5 (severe) for severity. Scores calculated as mean of item responses with higher scores indicating more severe or frequent symptoms.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm | Control
Number analyzed (Participants) | 39 | 21
Participants | 24 | 1

2. Primary Outcome: Number of Participants Reporting Elimination of Daily Troublesome Regurgitation Using a Validated Questionnaire for Assessment
Description: Elimination or clinically significant improvement in troublesome regurgitation refractory to PPIs as evaluated by the disease-specific and validated instrument, Reflux Disease Questionnaire (RDQ):12-item questionnaire assesses frequency and severity of heartburn (4 items measure frequency and severity of pain and burning behind breastbone), regurgitation (4 items measuring the frequency and severity of acid taste in mouth and movement of material upward from stomach), and dyspeptic complaints (4 items measure frequency and severity of pain or burning in upper stomach). Responses range from 0 (not present) to 5 (daily) for frequency and 0 (not present) to 5 (severe) for severity. Patient's score is calculated as the mean of item responses with higher scores indicating more severe or frequent symptoms. A frequency score of 3 or more and severity score of 2 or more for the regurgitation questions were required to meet the Montreal consensus criteria for troublesome regurgitation.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Groups:
- Control Arm: Participants taking standard dose PPI
Arm/Group | Treatment Arm | Control Arm
Number analyzed (Participants) | 30 | 18
Participants | 29 | 9

3. Secondary Outcome: Number of Participants With Complete PPI Discontinuation Assessed Using Validated Questionnaires and Participant-reported Discontinuation
Description: Elimination of daily bothersome GERD (Gastro Esophageal Reflux Disease) HRQL symptoms, using RDQ (Reflux Disease Questionnaire), RSI (Reflux Symptom Index) and as measured by complete discontinuation of PPI (Proton Pump Inhibitors) therapy at 6-month follow-up.
Time Frame: 6 Months
Measure: Count of Participants; unit: Participants
Groups:
- Control Arm: Participants taking maximum dose PPIs during Initial Study.
Arm/Group | Treatment Arm | Control Arm
Number analyzed (Participants) | 39 | 21
Participants | 35 | 0

4. Secondary Outcome: Number of Participants With Normalization of Esophageal Acid Exposure Assessed Using 48-hour pH Metry
Description: Assessment of esophageal acid exposure with normal defined as pH<4 in less than 5.3% total time exposure, using 48hr pH metry, with patients off PPIs for at least 7 days
Time Frame: 6 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm | Control Arm
Number analyzed (Participants) | 39 | 21
Participants | 21 | 11

5. Secondary Outcome: Number of Participants With Complete Healing or Reduction of Reflux Esophagitis, Assessed by EGD Using Los Angeles (LA) Grading
Description: Esophagitis graded using the LA grading system through endoscopic visualization. Data entered represents study participants with complete healing or reduction in reflux esophagitis compared to baseline results. Note that Control arm patients were assessed while on PPIs. LA grades are A, B, C, D, with A being the least severe. Grade D was an exclusion criteria. Normal has no associated grade.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Groups:
- Treatment Arm: Transoral incisionless esophagogastric fundoplication using the EsophyX system with SerosaFuse fasteners (EndoGastric Solutions, Inc., Redmond, WA, USA) and following TIF2.0 protocol.
  EsophyX System with SerosaFuse fasteners: Transoral Incisionless Fundoplication (TIF)/Transoral Incisionless Esophago-Gastric Fundoplication
- Control Arm: Patients taking standard daily dose of PPIs
Arm/Group | Treatment Arm | Control Arm
Number analyzed (Participants) | 20 | 13
Participants | 18 | 5

6. Other Pre Specified Outcome: Number of Participants With Elimination of Daily Troublesome Heartburn Assessed Using a Validated Questionnaire
Description: Elimination of daily bothersome heartburn as measured by GERD-HRQL (Gastro Esophageal Reflux Disease - Health-Related Quality of Life) questionnaire. GERD-HRQL is a validated questionnaire used to assess typical GERD symptoms by measuring 10 items on the visual analog scale ranging from 0 (no symptoms) to 5 (worst symptoms). A higher total GERD-HRQL score (range from 0 to 50) indicates more severe GERD.
  Note Control Arm patients are assessed while on standard daily dose of PPIs.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm | Control Arm
Number analyzed (Participants) | 31 | 16
Participants | 28 | 2

7. Post Hoc Outcome: Number of Participants With GERD Symptom Control Following TIF and Crossover TIF, Assessed by Validated Questionnaires (Primary Endpoint)
Description: Assess number of patients reporting global elimination of troublesome regurgitation and atypical symptoms using Reflux Disease Questionnaire (RDQ), a 12-item questionnaire to assess frequency and severity of heartburn (4 items measure frequency/severity of pain and burning behind breastbone), regurgitation (4 items measure frequency/severity of acid taste in mouth and movement of material upward from stomach), and dyspeptic complaints (4 items measure frequency and severity of pain or burning in upper stomach). Responses from 0 (not present) to 5 (daily) for frequency and 0 (not present) to 5 (severe) for severity, and Reflux Symptom Index (RSI), a 9-item questionnaire to assess atypical symptoms: hoarseness, throat clearing, excess throat mucus, dysphagia, cough. Scale for each item ranges from 0 (no problem) to 5 (severe), with max score of 45, normality threshold of ≤13. Scores calculated as mean of item responses with higher scores indicating more severe or frequent symptoms.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Groups:
- Control Arm: Patients who received Crossover TIF after 6-month initial study follow-up
Arm/Group | Treatment Arm | Control Arm
Number analyzed (Participants) | 39 | 20
Participants | 30 | 13

8. Post Hoc Outcome: Number of Participants Reporting Elimination of Troublesome Regurgitation Assessed Using a Validated Questionnaire (Primary Endpoint)
Description: Assessment of the number of patients reporting elimination of troublesome regurgitation using the validated Reflux Disease Questionnaire (RDQ), a 12-item questionnaire to assess frequency and severity of heartburn (4 items measure frequency/severity of pain and burning behind breastbone), regurgitation (4 items measure frequency/severity of acid taste in mouth and movement of material upward from stomach), and dyspeptic complaints (4 items measure frequency and severity of pain or burning in upper stomach). Responses from 0 (not present) to 5 (daily) for frequency and 0 (not present) to 5 (severe) for severity A frequency score of three or more and severity score of two or more for the regurgitation questions were required to meet the Montreal consensus criteria for troublesome regurgitation. The lower the score the better the outcome. (Crossover patients are 6-months post TIF.)
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm | Control Arm
Number analyzed (Participants) | 30 | 9
Participants | 28 | 6

9. Post Hoc Outcome: Number of Participants With Healing of Esophagitis After TIF and Crossover TIF (Secondary Endpoint)
Description: Assessment of number of participants reporting healed esophagitis after TIF using EGD and LA grading system. Treatment arm patients assessed at 12 month post TIF and Control arm patients are at 6 month post Crossover TIF (12 month post randomization). LA grading A, B, C, D, with A the least severe esophagitis. No grade listed is "Normal". Grade D is an exclusion criteria.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm | Control Arm
Number analyzed (Participants) | 19 | 13
Participants | 19 | 11

10. Post Hoc Outcome: Number of Participants With Normal Esophageal Acid Exposure Assessed Post-TIF and Post-Crossover TIF (Secondary Endpoint)
Description: as for outcome 4
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm | Control Arm
Number analyzed (Participants) | 38 | 21
Participants | 17 | 7

11. Post Hoc Outcome: Number of Participants Completely Off Daily PPIs Following TIF and Crossover TIF (Secondary Endpoint)
Description: Number of patients reporting complete cessation of daily PPI therapy at 12 months post TIF and 6 months post Crossover TIF. This is patient-reported.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm | Control Arm
Number analyzed (Participants) | 39 | 21
Participants | 32 | 15

12. Post Hoc Outcome: Number of Participants Reporting Elimination of Troublesome Regurgitation Assessed Using a Validated Questionnaire (Primary Endpoint)
Description: Assessment of the number of patients reporting elimination of troublesome regurgitation using the validated Reflux Disease Questionnaire (RDQ), a 12-item questionnaire to assess frequency and severity of heartburn (4 items measure frequency/severity of pain and burning behind breastbone), regurgitation (4 items measure frequency/severity of acid taste in mouth and movement of material upward from stomach), and dyspeptic complaints (4 items measure frequency and severity of pain or burning in upper stomach). Responses from 0 (not present) to 5 (daily) for frequency and 0 (not present) to 5 (severe) for severity. A frequency score of three or more and severity score of two or more for the regurgitation questions were required to meet the Montreal consensus criteria for troublesome regurgitation. The cohort of patients reported includes Treatment arm patients and Crossover patients combined as one group. Crossover patients included in the cohort are 30 months post TIF.
Time Frame: 36 months
Population: Extended Follow-up Phase will place all patients into one cohort, combining Treatment and Control arm patients. All become "Treatment" patients so Control arm number of participants becomes 0.
Measure: Count of Participants; unit: Participants
Groups:
- Treatment Arm: Transoral incisionless esophagogastric fundoplication using the EsophyX system with SerosaFuse fasteners (EndoGastric Solutions, Inc., Redmond, WA, USA) and following TIF2.0 protocol.
  EsophyX System with SerosaFuse fasteners: Transoral Incisionless Fundoplication (TIF)/Transoral Incisionless Esophago-Gastric Fundoplication
  NOTE: This Arm now includes Control arm patients, making one cohort of patients for the Extended Follow up Phase of the study.
- Control Arm: Patients who received Crossover TIF after 6-month initial study follow-up. NOTE: These patients will be added to the Treatment arm patients to become one cohort of patients for Extended Follow-up Phase.
Arm/Group | Treatment Arm | Control Arm
Number analyzed (Participants) | 41 | 0
Participants | 37 | 0

13. Post Hoc Outcome: Number of Study Participants Reporting Elimination of All Troublesome Atypical GERD Symptoms Assessed by Reflux Symptom Index (RSI) (Primary Endpoint)
Description: Assessment of atypical GERD symptoms (symptoms other than heartburn) using validated Reflux Symptom Index (RSI), a 9 item questionnaire with a 0-5 score for each, for a total of 45, and a normality threshold of ≤13. The lower the score the better the outcome.
  Control/Crossover arm patients included in this cohort are at 30 months post TIF.
Time Frame: 36 months
Population: Control/Crossover arm patients are included in the overall number of participants analyzed under the Treatment arm section, so Control arm number will be 0.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm | Control Arm
Number analyzed (Participants) | 48 | 0
Participants | 42 | 0

14. Post Hoc Outcome: Number of Participants With pH Normalization at 3-year Follow-up (Secondary Endpoint)
Description: Assessment of esophageal acid exposure with normal defined as pH<4 in less than 5.3% total time exposure, using 48hr pH metry, with patients off PPIs for at least 7 days.
  Note that patients originally in the Control/Crossover arm are at 30 months post TIF at this follow up period. Treatment and Control/Crossover patients are reported as a single cohort.
Time Frame: 36 months
Population: All patients are reported as one cohort, under the Treatment arm. Control arm number of participants analyzed will be 0. All are included in Overall Number in Treatment arm section.
Measure: Count of Participants; unit: Participants
Groups:
- Control Arm: Patients who received Crossover TIF after 6-month initial study follow-up. NOTE: These patients will be added to the Treatment arm patients to become one cohort of patients for Extended Follow-up Phase. The value entered in this section is 0.
Arm/Group | Treatment Arm | Control Arm
Number analyzed (Participants) | 40 | 0
Participants | 16 | 0

15. Post Hoc Outcome: Number of Participants With Complete Discontinuation of Daily PPI Therapy (Secondary Endpoint)
Description: Number of patients reporting complete cessation of daily PPI therapy at 36 months post TIF and 30 months post Crossover TIF combined into a single cohort.
Time Frame: 36 months
Population: Treatment and Control/Crossover patients are reported as a single cohort at this follow-up period.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm | Control Arm
Number analyzed (Participants) | 52 | 0
Participants | 37 | 0

16. Post Hoc Outcome: Number of Participants With Healed Esophagitis (Secondary Endpoint)
Description: Assessment of number of participants reporting healed esophagitis after TIF using EGD and LA grading system, LA grade A, B, C, D, with A meaning least severe esophagitis. No grade means normal.
  30 months post TIF for Crossover patients.
Time Frame: 36 months
Population: Control/Crossover patients have been added to the Treatment arm patients to make one combined cohort of patients. Control/Crossover patients are at 30 months post TIF.
Measure: Count of Participants; unit: Participants
Groups:
- Treatment Arm: Transoral incisionless esophagogastric fundoplication using the EsophyX system with SerosaFuse fasteners (EndoGastric Solutions, Inc., Redmond, WA, USA) and following TIF2.0 protocol.
  EsophyX System with SerosaFuse fasteners: Transoral Incisionless Fundoplication (TIF)/Transoral Incisionless Esophago-Gastric Fundoplication
  NOTE: This Arm now includes Treatment arm plus Control arm patients, making one cohort of patients for the Extended Follow up Phase of the study.
Arm/Group | Treatment Arm | Control Arm
Number analyzed (Participants) | 22 | 0
Participants | 19 | 0

17. Post Hoc Outcome: Number of Patients Satisfied With Their Current Health Condition (Secondary Endpoint)
Description: Satisfaction with current health condition OFF PPIs is reported as part of the GERD health-related quality of life questionnaire (GERD-HRQL), with 3 possible answers: satisfied, neutral or dissatisfied.
Time Frame: 36 months
Population: All patients included in one cohort, entered in the treatment arm section
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm | Control Arm
Number analyzed (Participants) | 43 | 0
Participants | 35 | 0

18. Post Hoc Outcome: Number of Participants With Elimination of Daily Troublesome Regurgitation (Primary Endpoint)
Description: Number of patients reporting elimination of troublesome regurgitation using the validated Reflux Disease Questionnaire (RDQ), a 12-item questionnaire to assess frequency and severity of heartburn (4 items measure frequency/severity of pain and burning behind breastbone), regurgitation (4 items measuring frequency/severity of acid taste in mouth and movement of material upward from stomach), and dyspeptic complaints (4 items measure frequency/severity of pain or burning in upper stomach). 9 response options range from 0 (not present) to 5 (daily) for frequency and 0 (not present) to 5 (severe) for severity. Each patient's score is calculated as the mean of item responses, with higher scores indicating more frequent and/or severe symptoms. Cohort of patients reported at this time period includes Treatment arm patients and Control/Crossover patients combined as 1 group. Control/Crossover patients included in cohort are at 54 months post TIF.
Time Frame: 60 months
Population: There were 44 patients available for follow up at 5 years post TIF. 43 were analyzed for regurgitation.
  Treatment and Control/Crossover patients were combined into one cohort, shown in Treatment arm. Control arm value is 0. Control/crossover patients are at 54 months post TIF.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm | Control Arm
Number analyzed (Participants) | 43 | 0
Participants | 37 | 0

19. Post Hoc Outcome: Number of Patients With Elimination of Troublesome Atypical GERD Symptoms (Primary Endpoint)
Description: Number of patients with elimination of troublesome GERD symptoms using Reflux Symptom Index (RSI), a 9-item validated questionnaire to measure atypical GERD symptoms such as hoarseness, throat clearing, excess throat mucus, dysphagia, and cough. The scale for each individual item ranges from 0 (no problem) to 5 (severe problem), with a maximum total score of 45 and a normality threshold of ≤13. The lower the score, the better the outcome.
Time Frame: 60 months
Population: Control/crossover patients are included in overall number of patients analyzed and entered in Treatment arm section to make one cohort. Crossover patients are at 54 month post TIF follow up.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm | Control Arm
Number analyzed (Participants) | 39 | 0
Participants | 31 | 0

20. Post Hoc Outcome: Number of Patients Reporting Complete Cessation of Daily PPIs (Secondary Endpoint)
Description: Number of participants with complete cessation of daily PPI use, self-reported by patient at 60 month follow-up. (54 months for Control/crossover patients). Note: all patients were on daily PPIs at screening (100%).
Time Frame: 60 months
Population: One cohort of patients entered as Overall number of Participants Analyzed, in Treatment arm section. Includes all available Control/crossover patients at 54 month post TIF follow up.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm | Control Arm
Number analyzed (Participants) | 44 | 0
Participants | 20 | 0

21. Post Hoc Outcome: Number of Participants Satisfied With Their Current Health Condition (Secondary Endpoint)
Description: Satisfaction with current health condition OFF PPIs is reported as part of the GERD health-related quality of life questionnaire (GERD-HRQL), with 3 possible answers: satisfied, neutral or dissatisfied. 60 months post TIF, 54 months post Crossover.
Time Frame: 60 months
Population: Overall Number of Participants Analyzed entered in Treatment arm includes all Control/crossover arm patients available for follow up. Control/crossover patients are at 54 month post-TIF follow up.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm | Control Arm
Number analyzed (Participants) | 44 | 0
Participants | 31 | 0

22. Post Hoc Outcome: Number of Participants Undergoing Reoperation Post-TIF (Secondary Endpoint)
Description: Reoperations completed post TIF by the end of 60 month (54 months post Crossover) follow up. These included 2 Laparoscopic Nissen fundoplications and 1 Dor fundoplication, completed without difficulty. This number includes the two reoperations reported and included in number of participants analyzed, at 36 month follow up.
Time Frame: 60 months
Population: All participants are included in the Overall Number of Participants Analyzed, under the Treatment arm section; reported as 1 cohort.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm | Control Arm
Number analyzed (Participants) | 60 | 0
Participants | 3 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over a period of 6 months
Arm/Group | Treatment Arm | Control
All-Cause Mortality (participants affected / at risk) | 0/41 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/24
Other Adverse Events (participants affected / at risk) | 2/41 | 0/24
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Arm (N=41) | Control (N=24)
Post operative TIF procedure (Gastrointestinal disorders) | 1 (1) | 0 (0) — Overnight hospital stay at Investigator discretion, due to post-op nausea and dizziness related to the TIF procedure.
Post operative TIF procedure (General disorders) | 1 (1) | 0 (0) — Overnight hospital stay due to allergic reaction to pain medication given for TIF post-op pain.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No